CLINICAL TRIAL: NCT07083739
Title: Phase II Clinical Trial on the Safety and Efficacy of TQB3473 Tablets in the Treatment of Persistent or Chronic Primary Immune Thrombocytopenia (ITP) in Adults
Brief Title: A Study on the Safety and Efficacy of TQB3473 Tablets in the Treatment of Persistent or Chronic Primary Immune Thrombocytopenia (ITP) in Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3473-II-01
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3473 Tablets (Experimental): TQB3473 Tablets 600 mg orally once daily for 24 consecutive weeks.
  Interventions: Drug: TQB3473 Tablets

INTERVENTIONS:
Drug: TQB3473 Tablets — TQB3473 tablet is a selective Spleen tyrosine kinase (Syk) inhibitor.

SUMMARY:
This study is an extension of the TQB3473-III-01 study, aimed at evaluating the safety and efficacy of TQB3473 tablets in adult patients with persistent or chronic ITP who have received at least one ITP standard treatment that is ineffective or has recurred after treatment. This is a single arm, open label, multi cohort, multi center Phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 :

* Voluntarily participate in this study with signed informed consent form (ICF) and demonstrated good compliance.
* Age ≥18 years (calculated from the date of ICF signing); no gender restrictions; Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Clinically stable condition with WHO bleeding scale score 0-1, and investigator assessment indicates no need for emergency treatment within the next 2 weeks.
* No increase in the type, dosage, or frequency of concomitant ITP medications compared to the TQB3473-III-01 study regimen.
* Previous participation in the TQB3473-III-01 study with either: Sustained platelet count <30×10⁹/L during the 12-week pre-randomization period (<50×10⁹/L if emergency treatment was received), or completion of 24-week double-blind treatment with investigator-confirmed benefit-risk assessment favoring continued therapy.
* Adequate major organ function as defined by protocol criteria.
* For women of childbearing potential: Must agree to use highly effective contraception from screening through 6 months after treatment completion and refrain from oocyte donation for reproductive purposes during this period; must not be breastfeeding with negative serum/urine pregnancy test within 7 days prior to enrollment. For male participants with fertile partners: Must agree to use effective contraception during the study and for 6 months thereafter.

Cohort 2 ：

* Subjects voluntarily participate in this study upon signing the Informed Consent Form (ICF) with demonstrated compliance.
* Age ≥ 18 years (calculated from signing date of ICF); No gender restrictions; ECOG performance status score 0-1.
* Confirmed diagnosis of primary ITP >3 months prior to enrollment.
* Clinically stable condition with WHO bleeding score 0-1, no major bleeding episodes within 4 weeks pre-randomization, and investigators confirm no anticipated need for emergency treatment within 2 weeks.
* Meeting all platelet criteria: Mean platelet count <30×10⁹/L (no single value >35×10⁹/L) from ≥2 independent measurements (≥3 days apart) within 7 days pre-enrollment Confirmed platelet count <30×10⁹/L within 24 hours before enrollment.
* Documented failure or relapse after ≥1 prior standard ITP therapy.
* Adequate function of major organs per protocol definitions.
* Permitted ≤1 concurrent ITP treatment (any class), provided: Stable dose maintained for ≥4 weeks prior to enrollment (≥2 weeks for corticosteroids)
* For women of childbearing potential: Must agree to use highly effective contraception from screening through 6 months after treatment completion and refrain from oocyte donation for reproductive purposes during this period; must not be breastfeeding with negative serum/urine pregnancy test within 7 days prior to enrollment. For male participants with fertile partners: Must agree to use effective contraception during the study and for 6 months thereafter.

Exclusion Criteria:

* Cohort 1 :

  1. Due to reasons other than lack of efficacy, receiving TQB3473-III-01 study treatment for less than 12 weeks.
  2. Hepatitis B Virus (HBV) DNA or Hepatitis C Virus (HCV) RNA detection values exceeding the upper limit of normal or decompensated cirrhosis
  3. Previous intracranial hemorrhage or severe bleeding of other important organs (≥ CTC AE grade 3), or symptomatic gastrointestinal bleeding (such as vomiting blood, black stool, etc., except for asymptomatic and asymptomatic "occult blood test positive" and hemorrhoids) within the 6 months before enrollment.
  4. Suffering from major cardiovascular and cerebrovascular diseases.
  5. There are multiple factors that can affect oral medication, such as inability to swallow, chronic diarrhea, and intestinal obstruction.
  6. Those who have received major surgical treatment, significant traumatic injury, or are expected to undergo major elective surgery during the study treatment period within the 4 weeks prior to enrollment
  7. Uncontrolled significant active infections (such as sepsis, pneumonia, or abscess), or severe infections within the 12 weeks prior to enrollment (resulting in hospitalization or requiring antibiotic treatment).
  8. Vaccination was administered within 8 weeks prior to enrollment, or planned during the study period.
  9. Received blood transfusions or blood products within 2 weeks prior to enrollment (excluding IVIg used for emergency treatment).
  10. Take strong CYP3A inhibitors or inducers (3 weeks for Forsythia suspensa) for 2 weeks or 5 half lives (whichever is longer) before enrollment.
  11. Long term/continuous treatment with drugs that affect platelet function (including but not limited to aspirin, clopidogrel, ticagrelor, NSAIDs, etc.) or anticoagulant therapy is required.
  12. Allergic constitution or history of severe allergies, or known allergies to the components of the investigational drug excipients.
  13. There are clear neurological or mental disorders, or serious psychological or mental abnormalities.
  14. Alcoholic or drug abusers.
  15. According to the researcher's perspective, other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that may increase the risks associated with participating in the study or interfere with the interpretation of the research results.
  16. It is estimated that the patient's compliance in participating in this clinical study is insufficient.

Cohort 2：

* There is evidence to suggest the presence of secondary causes of ITP in the subjects, or immune cell depletion of two or more lineages, such as Evans syndrome;
* Past or current presence of myelofibrosis, myelodysplastic syndrome, aplastic anemia, lymphoproliferative disorders, or other malignant hematological diseases.
* Have had or currently have malignant tumors within the past 3 years. The following two situations can be included in the group: other malignant tumors treated with a single surgery, achieving continuous 5-year disease-free survival (DFS); Cured cervical carcinoma in situ, non melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basement membrane)].
* HBV DNA or HCV RNA detection values exceeding the upper limit of normal or decompensated cirrhosis.
* Previous intracranial hemorrhage or severe (≥ Common Terminology Criteria (CTC) AE grade 3) bleeding of other important organs, or symptomatic gastrointestinal bleeding (such as vomiting blood, black stool, etc., except for asymptomatic and asymptomatic "occult blood test positive" and hemorrhoids) within the 6 months before enrollment.
* Suffering from major cardiovascular and cerebrovascular diseases.
* There are multiple factors that can affect oral medication, such as inability to swallow, active gastric ulcers, major gastrointestinal surgeries, chronic diarrhea, and intestinal obstruction.
* ITP related symptoms and treatment:

  * Received ITP emergency treatment within 2 weeks prior to enrollment;
  * Received platelet transfusion within 2 weeks prior to enrollment;
  * Received immunoglobulin or traditional Chinese medicine treatment within 2 weeks before enrollment;
  * Used rituximab or other anti-Cluster of Differentiation 20 (CD20) drugs within 14 weeks prior to enrollment;
  * Received splenectomy within 12 weeks prior to enrollment;
  * Individuals who have received glucocorticoids within the 2 weeks prior to enrollment, or have received thrombopoietin drugs (rhTPO, eltrombopag, hetrombopag, avatrombopag, romiplostim), immunomodulators (azathioprine, cyclosporine A, mycophenolate mofetil), chemotherapy drugs (decitabine, vinblastine), danazol, etc. within the 4 weeks prior to enrollment, except for those who meet the inclusion criteria 8 and are allowed to undergo concomitant treatment.
* Adverse reactions from previous treatments that have not recovered to ≤ CTCAE grade 1, as well as non clinically significant and asymptomatic laboratory abnormalities that have been determined by researchers to pose no safety risks, are excluded.
* Patients who have received major surgical treatment, significant traumatic injury, or are expected to undergo major elective surgery during the study treatment period within the 4 weeks prior to enrollment (major surgery is defined as surgery at level 3 or above in the National Surgical Classification Catalogue 2022 edition).
* Vaccination was administered within 8 weeks prior to enrollment, or planned during the study period.
* Uncontrolled significant active infections (such as sepsis, pneumonia, or abscess), or severe infections within the 12 weeks prior to enrollment (resulting in hospitalization or requiring antibiotic treatment).
* Received blood transfusions or blood products within 2 weeks prior to enrollment (excluding intravenous immunoglobulin (IVIg) used for emergency treatment).
* Take strong Cytochrome P450 3A (CYP3A) inhibitors or inducers (3 weeks for Forsythia suspensa) for 2 weeks or 5 half lives (whichever is longer) before enrollment.
* Participants who have participated in and used other clinical trial drugs within 4 weeks prior to enrollment.
* Long term/continuous treatment with drugs that affect platelet function (including but not limited to aspirin, clopidogrel, ticagrelor, NSAIDs, etc.) or anticoagulant therapy is required.
* Allergic constitution or history of severe allergies, or known allergies to the components of the investigational drug excipients.
* History of important organ transplantation or hematopoietic stem cell/bone marrow transplantation.
* History of immunodeficiency, including HIV positivity or other congenital immunodeficiency diseases.
* Individuals with epilepsy who require treatment.
* There are clear neurological or mental disorders, or serious psychological or mental abnormalities.
* Alcoholic or drug abusers.
* According to the researcher's perspective, other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that may increase the risks associated with participating in the study or interfere with the interpretation of the research results.
* It is estimated that the patient's compliance in participating in this clinical study is insufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Sustained response rate | Weeks 13-24
  During the last 12 weeks of treatment, at least 2 platelet counts were ≥50×10^9/L in three protocol-determined visits (excluding rescue treatment).

SECONDARY OUTCOMES:
Response rate at 12 weeks | Within 12 weeks of treatment
  ① The percentage of patients with platelet count ≥ 50×10^9/L at least once within 12 weeks of treatment (excluding emergency treatment). ② The percentage of subjects with a baseline platelet count of<15 × 10^9/L who have had at least one platelet count of ≥ 30×10^9/L within 12 weeks of treatment and an increase of ≥ 20 × 10^9/L from baseline (excluding emergency treatment);
Response rate at 24 weeks | Within 24 weeks of treatment
  * The percentage of patients with platelet count ≥ 50×10^9/L at least once within 24 weeks of treatment (excluding emergency treatment).
    * The percentage of subjects with a baseline platelet count of<15 × 10^9/L who have had at least one platelet count of ≥ 30×10^9/L within 24 weeks of treatment and an increase of ≥ 20 × 10^9/L from baseline (excluding emergency treatment); ③ The percentage of subjects with platelet counts at least twice the baseline level and ≥30×10^9/L for at least two consecutive measurements within 24 weeks of treatment (excluding rescue treatment).
Time to Onset | Within 24 weeks of treatment
  The time from the initiation of treatment to the first platelet count ≥50×10^9/L
The cumulative duration of platelet count ≥ 50 × 10^9/L within 24 weeks of treatment | Within 24 weeks of treatment
  The cumulative duration of platelet count ≥ 50 × 10^9/L within 24 weeks of treatment.
The proportion of subjects who receive rescue treatment | Within 24 weeks of treatment
  The proportion of subjects who receive rescue treatment aimed to increase platelet counts within 24 weeks of treatment.
The incidence and severity of bleeding events | Within 24 weeks of treatment
  The incidence and severity of bleeding events evaluated according to the World Health Organization (WHO) bleeding scoring criteria within 24 weeks of treatment.
The change of concomitant therapy | Within 24 weeks of treatment
  The proportion of subjects who reduce or discontinue concomitant ITP treatments within 24 weeks of treatment.
Improvement in Quality of Life Score | Within 24 weeks of treatment
  Conduct a comprehensive evaluation of the physical condition of the subjects, and the higher the score, the better the subject's condition.
The incidence and severity of adverse events (AE) and serious adverse events (SAE), as well as abnormal laboratory test indicators. | Within 24 weeks of treatment
  The incidence and severity of adverse events (AE) and serious adverse events (SAE), as well as abnormal laboratory test indicators.
Area under the curve (0 to Infinity) after initial administration (AUC0-∞) | Within 24 weeks of treatment
  Main pharmacokinetic parameters, area under the curve (0 to Infinity) after initial administration (AUC0-∞)
Maximum plasma concentration (Cmax) after initial administration | Within 24 weeks of treatment
  Maximum plasma concentration (Cmax) after initial administration.
Elimination Half-Life（t1/2）after initial administration | Within 24 weeks of treatment
  Elimination Half-Life（t1/2）after initial administration.
Apparent clearance（CL/F）after initial administration | Within 24 weeks of treatment
  Apparent clearance（CL/F）after initial administration.
Apparent Volume of Distribution (Terminal Phase)（Vz/F）after initial administration | Within 24 weeks of treatment
  Apparent Volume of Distribution (Terminal Phase)（Vz/F）after initial administration.
Terminal elimination Rate Constant (λz) after initial administration | Within 24 weeks of treatment
  Terminal elimination Rate Constant (λz) after initial administration.
Area under the curve (0 to 24 hours) after multiple administration (AUC0-24h) | Within 24 weeks of treatment
  Area under the curve (0 to 24 hours) after multiple administration (AUC0-24h).
Area under the curve (0 to Infinity) after multiple administration (AUC0-∞) | Within 24 weeks of treatment
  Area under the curve (0 to Infinity) after multiple administration (AUC0-∞).
Minimum steady-state concentration (Css-min) after multiple administration | Within 24 weeks of treatment
  Minimum steady-state concentration (Css-min) after multiple administration.
Maximum steady-state concentration (Css-max) after multiple administration | Within 24 weeks of treatment
  Maximum steady-state concentration (Css-max) after multiple administration.
Average Steady-State Concentration (Css-avg) after multiple administration | Within 24 weeks of treatment
  Average Steady-State Concentration (Css-avg) after multiple administration.
Elimination Half-Life (t1/2) after multiple administration | Within 24 weeks of treatment
  Elimination Half-Life (t1/2) after multiple administration.
Apparent Clearance (CL/F) after multiple administration | Within 24 weeks of treatment
  Apparent Clearance (CL/F) after multiple administration.
Apparent volume of distribution (Steady State) after multiple administration (Vss/F) | Within 24 weeks of treatment
  Apparent volume of distribution (Steady State) after multiple administration (Vss/F).
Terminal Elimination Rate Constant (λz) after multiple administration | Within 24 weeks of treatment
  Terminal Elimination Rate Constant (λz) after multiple administration.
Accumulation ratio constant (Rac) after multiple administration | Within 24 weeks of treatment
  Accumulation ratio constant (Rac) after multiple administration.
Degree of fluctuation (DF) after multiple administration | Within 24 weeks of treatment
  Degree of fluctuation (DF) after multiple administration.

CONTACTS AND LOCATIONS:
Locations (51):
- China (51):
  - The first affiliated hospital of ustc anhui provincial hospital, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Nanshan People's Hospital, Shenzhen, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei University / School of Clinical Medicine, Baoding, Hebei
  - Affiliated Hospital of ChengDe Medical University, Chengde, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University of science and technology, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First People's Hospital of Ping Ding Shan, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Shenjing Hospital Of China Medical University, Shenyang, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Xijing Hospital, Xi'an, Shaanxi
  - Xi'an No.3 Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Central Hospital, Jinan, Shandong
  - Linyi Central Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital (Affiliated Yantai Yuhuangding Hospital of Qingdao University), Yantai, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Qingpu Branch, Shanghai, Shanghai Municipality
  - Heping Hospital affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Kunming Medical University Second Affiliated Hospital, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang